CLINICAL TRIAL: NCT01054924
Title: Clinical Study to Assess the Performance of the Invendo C20 Colonoscope System in Persons Undergoing Colorectal Cancer Screening at Average Risk for CRC
Brief Title: Performance Study of the Invendo C20 Colonoscope System in Colorectal Cancer Screening
Status: Completed | Type: Observational
Sponsor: Invendo Medical GmbH (Industry)
Other Study IDs: INV2009-01
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- U.S. CRC screening population

SUMMARY:
The purpose of the study is to evaluate efficacy (i.e. reaching the cecum) and safety of the Invendo C20 Colonoscopy System

ELIGIBILITY:
Inclusion Criteria:

1. Screenees, i.e. asymptomatic persons willing to undergo screening colonoscopy, at average risk for colorectal cancer
2. Age between 50-75 years
3. Signed informed consent

Exclusion Criteria:

1. Family or personal history of colorectal neoplasia including familial adenomatous polyposis (FAP) or hereditary non-polyposis colorectal cancer
2. Prior colonoscopy within preceding 10 years
3. A suspected diagnosis of inflammatory bowel disease, bowel obstruction, acute diverticulitis, known severe diverticulosis or any known large bowel disease
4. Clinically significant cardiovascular or pulmonary diseases
5. Gastrointestinal-tract related symptoms, complaints or diseases suggesting performance of colonoscopy (no screening cases)
6. Cancer or other life threatening diseases or significant chronic conditions
7. Blood clotting disorders and /or anti-coagulant therapy including aspirin within the last 7 days
8. Known pregnancy or positive screening pregnancy tests
9. Previous abdominal surgery except for uncomplicated cholecystectomy, appendectomy or minor pelvic surgery (e.g. hernia repair, oophorectomy)
10. Morbid obesity (BMI > 40)
11. Clinically significant abnormal screening laboratory findings
12. Clinically significant abnormal screening ECG findings
13. Drug abuse or alcoholism
14. Inability of the screenee to adequately communicate
15. Screenees under custodial care
16. Participation in a clinical study within the last 30 days

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic persons fulfilling U.S. screening criteria for colorectal cancer of age of 50-75 years
Sampling Method: Non-Probability Sample
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Roesch, Prof., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Nicolas Hoepffner, MD, Principal Investigator — Centrum Gastroenterologie Bethanien, Frankfurt; Douglas K. Rex, Prof., Principal Investigator — Indiana University Hospital
Locations (2):
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Centrum Gastroenterologie Bethanien, Frankfurt am Main, Hesse